CLINICAL TRIAL: NCT04174742
Title: Self-Reported Pain and Nadir White Blood Cell/Absolute Neutrophil Count in Women 45 and Under Compared to Older Women Receiving Pegfilgrastim (or Biosimilar Substitution) While Undergoing Chemotherapy for Non-Metastatic Breast Cancer
Brief Title: Self Reported Pain in Women While Undergoing Treatment for Non-metastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00081356; Pro00037721 (Other: Advarra IRB); LCI-BRE-GCSF-001 (Other: Atrium Health)
Record Dates: First submitted 2019-10-31; First posted 2019-11-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast; Breast Cancer
Keywords: Pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — pegfilgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A: Subjects 45 years of age or younger
  Interventions: Drug: pegfilgrastim
- B: Subjects over 45 years of age
  Interventions: Drug: pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim — It works by increasing neutrophil migration to counteract cytotoxicity. It is commonly administered to patients receiving chemotherapy for breast cancer treatment. It has been shown to significantly reduce the incidence of neutropenic fever, although without statistically significant impact on overall survival.

SUMMARY:
The overall purpose of this study is to investigate whether younger subjects report pain with pegfilgrastim (or biosimilar substitution) more often and/or at higher levels (greater intensity) than older subjects.This study will be carried out throughout the course of your chemotherapy treatment, which will be prescribed by your study doctor. Participation in this study will not affect your cancer treatment.

DETAILED DESCRIPTION:
This study will measure pain using ESAS self-reported pain scores over the course of one week following each dose of pegfilgrastim (or biosimilar substitution). At the end of that week, blood will be drawn from each subject to directly measure the WBC/ANC, which can then be compared to self-reported pain and evaluated for any correlation. Finally, subjects will be divided into two groups by age: 45 years or younger, and over 45 to look for any differences in pain or WBC/ANC measurements based on age.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent
3. Female
4. Histological or cytological confirmation of invasive breast cancer.
5. Planned to undergo adjuvant or neoadjuvant chemotherapy treatment for invasive breast cancer AND pegfilgrastim (or biosimilar substitution) treatment for neutropenic prophylaxis.
6. Ability to read and understand the English and/or Spanish language
7. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

1. Uncontrolled intercurrent illness/medical condition or psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator
2. Have previously received chemotherapy or radiation other than the first cycle of the planned adjuvant or neoadjuvant chemotherapy as indicated in Inclusion #5
3. Taking chronic narcotics, as determined by treating physician
4. Diagnosis of distant metastatic breast cancer
5. Diagnosis of a chronic pain syndrome (e.g. fibromyalgia, severe osteoarthritis, etc.)
6. A baseline ESAS pain score of greater than 8.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients undergoing neoadjuvant or adjuvant chemotherapy for breast cancer who will receive pegfilgrastim (or biosimilar substitution) during their treatment.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2041-01 (Estimated); Study Completion 2041-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of pain | approx 7 months
  investigate whether younger patients report pegfilgrastim (or biosimilar substitution)-induced pain with greater frequency than older patients.

SECONDARY OUTCOMES:
Intensity of pain | approx 7 months
  investigate whether younger patients report pegfilgrastim (or biosimilar substitution)-induced pain at a higher intensity than older patients.
White Blood Cell/Absolute Neutrophil Count (WBC/ANC) | On day 7 of each pegfilgrastim or biosimilar substitution cycle (28 day cycle, approx 4-6 cycles) through study completion (one week after last administration of pegfilgrastim or biosimilar substitution)
  compare WBC/ANC count nadir between younger and older patients receiving pegfilgrastim (or biosimilar substitution).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fisher, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina